CLINICAL TRIAL: NCT03022578
Title: Phase II Study of Laser Interstitial Thermal Therapy (LITT) in Recurrent Glioblastoma
Brief Title: Laser Interstitial Thermal Therapy and Lomustine in Treating Patients With Recurrent Glioblastoma or Anaplastic Astrocytoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0443; NCI-2018-01286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0443 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: IDH Family Wildtype; Recurrent Anaplastic Astrocytoma; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (LITT, lomustine) (Experimental): Patients undergo LITT at baseline and receive lomustine PO on day 1. Treatment with lomustine repeats every 42 days for up to 6 cycles in the absence of disease progression or unaccepted toxicity.
  Interventions: Procedure: Laser Interstitial Thermal Therapy; Drug: Lomustine

INTERVENTIONS:
Procedure: Laser Interstitial Thermal Therapy — Undergo LITT
  Other Names: LITT
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N''-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017

SUMMARY:
This phase II trial studies how well laser interstitial thermal therapy and lomustine work in treating patients with glioblastoma or anaplastic astrocytoma that has come back. Using laser to heat the tumor cells may help to kill them. Drugs used in chemotherapy, such as lomustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving laser interstitial thermal therapy and lomustine may work better in treating patients with glioblastoma or anaplastic astrocytoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the disease control rate at 6 months in patients with recurrent glioblastoma or isocitrate dehydrogenase (IDH)-wildtype anaplastic astrocytoma treated with Laser Interstitial Thermal Therapy (LITT) at recurrence, followed by salvage chemotherapy.

SECONDARY OBJECTIVES:

I. Estimate overall survival (OS) of patients with recurrent glioblastoma, or isocitrate dehydrogenase (IDH)-wildtype anaplastic astrocytoma treated with LITT at tumor recurrence, followed by salvage chemotherapy.

II. Estimate time to progression (TTP) of patients with recurrent glioblastoma, or isocitrate dehydrogenase (IDH)-wildtype anaplastic astrocytoma that are treated with LITT at tumor recurrence, followed by salvage chemotherapy.

III. Analyze volumetric data consisting of thermal damage threshold lines and overall tumor volume to determine any role of 'extent of ablation' in outcomes (OS and/or TTP).

IV. Characterize the safety profile of LITT followed by treatment with lomustine chemotherapy in the recurrent disease setting, using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

V. Assess the long-term steroid requirements following LITT, compared to historical controls.

VI. Determine the radiographic evolution of LITT-treated glioblastoma over time, using conventional magnetic resonance imaging (MRI) (T1 pre and post-contrast images, T2-weighted images [T2WI], fluid attenuating inversion recovery [FLAIR] images) and advanced brain tumor imaging (ABTI) [magnetic resonance (MR) perfusion [dynamic susceptibility contrast (DSC), dynamic contrast enhancement (DCE) and arterial spin labeling (ASL)], MR-diffusion, and MR spectroscopy), to include quantitative tumor metrics (volumetric extent of ablation and Response Assessment in Neuro-Oncology [RANO] criteria).

VII. Analyze health care utilization as measured by length of hospital stay following LITT (including inpatient rehabilitation care).

VIII. Evaluate patients' functional status (using the Karnofsky performance score [KPS] and the occurrence of symptoms [using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT[English])] self-reporting tool), and correlate to disease progression and tolerance to treatment.

EXPLORATORY OBJECTIVES:

I. Identify correlative tumor and peripheral blood molecular markers that impact outcomes, etc, and identify inflammatory/immunologic markers to assess neoantigen expression, etc, if sufficient tissue is available.

II. Identify and characterize changes in tumor tissue following LITT, by analyzing and comparing pre- and post-procedure tissue samples, if sufficient tissue is available.

OUTLINE:

Patients undergo LITT at baseline and receive lomustine orally (PO) on day 1. Treatment with lomustine repeats every 42 days for up to 6 cycles in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-proven, recurrent supratentorial grade IV glioblastoma (or grade III IDH-wildtype anaplastic astrocytoma), for which a complete surgical resection is unsafe due to location, shape, or size of the tumor. Diagnosis of recurrence will be established by biopsy and frozen section immediately prior to initiating LITT procedure. If findings on frozen section are not consistent with recurrence (glioblastoma or recurrent IDH-wildtype anaplastic astrocytoma), decision to proceed with LITT procedure will be at the discretion of the neurosurgeon (only patients with histologically-proven recurrent tumor will be evaluable for efficacy).
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information. Patients must be registered prior to treatment on study.
* Patients must have a Karnofsky performance score (KPS) > 60.
* Patients must have received standard of care therapy with chemoradiation with temozolomide followed by adjuvant chemotherapy with temozolomide. Patients may have received one additional chemotherapy regimen (other than lomustine) in addition to adjuvant temozolomide prior to study entry (patients at either first or second recurrence are eligible).
* In the context of this clinical trial, a lesion suitable for LITT is single, enhancing, supratentorial, at least 2 cm from inner table of skull over the hemispheric convexity, and > 1 cm, but < 4 cm in cross-sectional dimension, including thalamic tumor (=< 3 cm).
* Patients must have stable cardiovascular, neurovascular and neurological status, and be considered surgical candidates, as determined by any relevant pre-operative assessments, at the neurosurgeon's discretion.
* Patients must not be receiving concurrent anti-tumor treatment and must have recovered from toxicity of prior treatment. Minimum interval required: 1) > 6 weeks following nitrosourea chemotherapy; 2) > 4 weeks after recovering from any non-nitrosourea drug or systemic investigational agent; 3) > 2 weeks after receiving any non-cytotoxic anti-tumor drug; 4) > 4 weeks after receiving radiation therapy (> 12 weeks following upfront concurrent chemoradiation); 5) > 2 weeks following Optune device use.
* Patients must not have previously undergone an intracranial LITT procedure.
* White blood cell (WBC) > 3,000/ul (performed within 14 days (+ 3 working days) prior to registration)
* Absolute neutrophil count (ANC) > 1,500/mm^3 (performed within 14 days (+ 3 working days) prior to registration)
* Platelet count of > 100,000/mm^3 (may be reached by transfusion) (performed within 14 days (+ 3 working days) prior to registration)
* Hemoglobin > 10 gm/dl (may be reached by transfusion) (performed within 14 days (+ 3 working days) prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin < 2 times upper limit of normal (ULN) (performed within 14 days (+ 3 working days) prior to registration)
* Creatinine < 1.5 mg/dL (performed within 14 days (+ 3 working days) prior to registration)
* Women of childbearing potential must have a negative B-Human chorionic gonadotropin (HCG) documented within 7 days prior to registration and must agree to practice adequate contraception as defined below. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), includes any female who has had:

  * A hysterectomy
  * A bilateral oophorectomy
  * A bilateral tubal ligation
  * Is post-menopausal: Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L).
* Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT.
* Childbearing potential includes any female who has had a negative serum pregnancy test within 7 days of study registration, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

  * Complete abstinence from sexual intercourse for 14 days before starting treatment, through the treatment, and for at least 1 month after the last dose of temozolomide
  * Oral contraceptive, either combined or progestogen alone. A second barrier method is required during the first month of treatment with oral contraceptives
  * Injectable progesterone
  * Implants of levonorgestrel
  * Estrogenic vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
  * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
  * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository). Female participants who are lactating should discontinue nursing prior to the first dose of temozolomide and should refrain from nursing throughout the treatment period and for 42 days following the last dose of lomustine.

Exclusion Criteria:

* Patients must not have received prior treatment with bevacizumab.
* Patients must not have had prior treatment of glioblastoma with stereotactic radiosurgery, brachytherapy, or carmustine-impregnated wafers (Gliadel).
* Patients must not have symptoms attributed to mass effect of the tumor (despite corticosteroid treatment) that would be better treated with debulking surgery, or wherein surgical debulking in the first 30 days following LITT procedure would be anticipated for symptom management.
* Patients unable to undergo MRI are not eligible.
* Patients with progression of multifocal tumors or tumors involving the posterior fossa (brainstem and cerebellum) will be excluded, as will patients where the anticipated treatment margin will be within 5 mm of critical intracranial structures (e.g., primary branches of cerebral vessels, dural sinuses, hypophysis or cranial nerves).
* Patients may not have undergone previous treatment with lomustine.
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients must not have active infection or serious intercurrent medical illness.
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception.
* Patients must not have uncontrolled hypertension (systolic >180 mm hg or diastolic > 100 mg Hg), angina pectoris, cardiac dysrhythmia, or recent (within 6 weeks) intracranial hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J O'Brien, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 Participants signed consent, 3 participants inevaluable due to screen failure
Period: Overall Study
Arm/Group | Treatment (LITT, Lomustine)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 57 [37 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate at 6 Months
Description: Stable Disease per RANO occurs if the patient does not qualify for response or progression and requires stable non enhancing lesions, same/lower dose of corticosteroids, and clinical stability.
  Complete Response per RANO requires complete disappearance of all enhancing measurable and nonmeasurable disease for at least 4 weeks; no new lesions; and stable/improved nonenhancing lesions, off corticosteroids (or on physiologic replacement dose) and clinical improvement/stability. Partial Response per RANO requires ≥50% decrease of enhancing lesions compared with baseline, sustained for at least 4 weeks; no progression of nonmeasurable disease; no new lesions; stable/improved nonenhancing lesions, same/lower dose of corticosteroids not greater than the dose at time of the baseline scan and clinically improved/stable.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
Participants
  Progression Disease | 2
  Partial Response | 1
  Non Evaluable | 1

2. Secondary Outcome: Time to Progression (TTP)
Description: Progression disease per the Response Assessment in Neuro-Oncology (RANO) is defined by any of the following: ≥25% increase in the sum of the products of perpendicular diameters of enhancing lesions (compared with baseline if no decrease) on stable or increasing doses of corticosteroids; a significant increase in T2/FLAIR nonenhancing lesions on stable or increasing doses of corticosteroids compared with the baseline scan or the best response after initiation of therapy, not due to comorbid events; the appearance of any new lesions; clear progression of nonmeasurable lesions; or definite clinical deterioration not attributable to other causes apart from the tumor or to a decrease in the corticosteroid dose.
Time Frame: From date of enrollment in study to the date of first observation of progressive disease, death due to disease (event), or early discontinuation of treatment, approximately 3 years 3 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
weeks | 30 [1 to 63]

3. Secondary Outcome: Long-term Steroid Requirements
Description: Will be summarized by frequency tables.
Time Frame: Up to 4 years
Population: Data were not collected.
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 0

4. Secondary Outcome: MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) Data
Description: Will summarize the MDASI-BT at each time point using descriptive statistics and evaluate the change of MDASI-BT over time and its correlation with response and/or treatment tolerance using linear mixed models, where random effects will be used to account for within-subject correlations.
Time Frame: at baseline, after procedure, and with every imaging visit thereafter, up to 4 years
Population: Data were not collected.
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Incidence of Toxicity (Significant Hemorrhage or Brain Herniation) Documented on Imaging
Description: Safety and toxicity of LITT by determination of adverse events and surgical complications within 2 weeks of the procedure, plus an additional 4 weeks (to account for potential delayed inflammatory changes and initiation of subsequent treatment). Safety for LITT procedure will be defined as the absence of severe clinical toxicity as determined by the CTCAE version 4.0, within 6 weeks of the procedure, and/or absence of acute events (ie, significant hemorrhage or brain herniation) documented on imaging. Severe toxicity will also be defined as a drop of 20 points or more in KPS and not amenable to corticosteroids, and likely attributable to the procedure, or symptomatic hemorrhage, increased brain edema resulting in herniation/impending herniation, and/or significant neurologic decline not amenable to corticosteroids. Safety and toxicity will be reassessed again throughout the duration of the study.
Time Frame: approximately 3 years 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is the time from initial tumor diagnosis (definitive surgical resection or biopsy) to death from any cause. Will be estimated using the Kaplan-Meier method and the comparison between or among patient's characteristic groups will be evaluated by log-rank test. The Cox regression model may be applied to assess the effect of covariates of interest on OS.
Time Frame: approximately 3 years 3 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
weeks | 69 [9 to 164]

7. Secondary Outcome: Length of Hospital Stay Following LITT
Description: The length of hospital stay in days, weeks or months. Length of Hospital stay was summarized by using standard descriptive statistics, such as mean, standard deviation, median, and range for continuous variables, frequency and proportion for categorical variables.
Time Frame: approximately 3 years 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 4
days | 3 [3 to 4]

8. Other Pre Specified Outcome: Biomarkers in Peripheral Blood and Tumor Tissue
Description: Will be summarized using standard descriptive statistics, such as mean, standard deviation, median, and range for continuous variables, frequency and proportion for categorical variables. Correlation will be assessed among continuous variables using Pearson or Spearman correlation coefficient, whichever is appropriate. Association between categorical variables will be examined by Chi-Squared test or Fisher's exact test when appropriate. Wilcoxon rank-sum test or Kruskal-Wallis test will be used to examine the difference on continuous variables between or among patient's characteristic groups.
Time Frame: Up to 4 years
Population: Data were not collected.
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Inflammatory/Immunologic Profile
Description: as for outcome 8
Time Frame: Up to 4 years
Population: Data were not collected.
Arm/Group | Treatment (LITT, Lomustine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from the start of treatment through 30 days after the last dose of treatment, approximately 3 years 3 months.
Arm/Group | Treatment (LITT, Lomustine)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (LITT, Lomustine) (N=4)
Muscle weakness right sided (Nervous system disorders) | 1
Paaresthesia (right arm numbnes) (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Dysphasia (aphasia) (Nervous system disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (LITT, Lomustine) (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dysphasia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Muscle weakness right-sided (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03022578/Prot_SAP_000.pdf